CLINICAL TRIAL: NCT01649726
Title: Comparison of Two Strategies to Realize Apnea Test for the Diagnostic of Brain Death in Potential Organ Donors (CPAPNEE STUDY)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CPAPNEE STUDY
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Alternative Method of Apnea Test

ARMS (2):
- Standard strategy (Other): Apnea test according to recommendations
  Interventions: Procedure: Apnea test - control
- CPAP strategy (Experimental): Apnea test with CPAP connection
  Interventions: Procedure: Apnea test - CPAP

INTERVENTIONS:
Procedure: Apnea test - control
  Arms: Standard strategy
Procedure: Apnea test - CPAP
  Arms: CPAP strategy

SUMMARY:
Clinical diagnostic of brain death requires a non-reactive coma, absence of brain stem reflex, and absence of spontaneous breathing. The confirmation of absence of spontaneous breathing is established the apnea test (according to the American Academy of Neurology's Guidelines). However this test may lead to complications (acute hypoxemia, ventilatory and cardiocirculatory disorders) and reduces significantly the number of lung transplants. Some data suggest modifying the apnea test : replace the ventilator switching off with continuous positive airway pressure (CPAP) use. These studies showed that this alternative method (CPAP) increased the level of lung harvest but they were not sufficient because these studies were monocentric, non randomized and with little patients,. That why the aim of the present study is to compare the standard strategy and CPAP strategy with a prospective, multicenter, randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Age : from 18 to 70 years
* Neurological signs evoking cerebral ischemia

Exclusion Criteria:

* Severe hypoxemia (PaO2/FiO2 < 200) with controlled ventilation (FiO2: 100%)
* Hypothermia < 36°C
* Obesity (BMI ≥ 40) with documented hypopnoea
* Intractable hypotension despite optimal filling and catecholamine doses > 1µg.Kg.min
* Patients with contraindication for organs harvesting.
* Documented chronic respiratory failure
* Progressive infectious acute respiratory disease
* Family opposition to subject's participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Eligibility to donor lung harvest

SECONDARY OUTCOMES:
Level of hypoxemia
Arterial blood gas after th apnea test
Rate of ventilatory disorder
Rate of cardiocirculatory disorder
Rate of apnea test interruption
Number of lung transplantation realization

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Angers University Hospital, Angers
  - Angoulême Hospital, Angoulême
  - Tours University Hospital, Chambray-lès-Tours
  - La Roche sur Yon Hospital, La Roche-sur-Yon
  - La Rochelle Hospital, La Rochelle
  - Limoges University Hospital, Limoges
  - Nantes University Hospital, Nantes
  - Nice University Hospital, Nice
  - Orléans Hospital, Orléans
  - Cochin University Hospital, Paris
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Saintes Hospital, Saintes